CLINICAL TRIAL: NCT01010217
Title: Three-arm Clinical Trial for Patients With Hematologic Malignancies and Mismatched Donors - Haploidentical, 1 Antigen Mismatch Related or Unrelated, and Matched Unrelated Donor (MUD)- Using a T-cell Replete Allograft and High-dose Post-transplant Cyclophosphamide
Brief Title: Mismatched Transplantation Using High-dose Post-transplant Cyclophosphamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0266; NCI-2011-03144 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Blood Stem Cell Transplant Failure; Leukemia; Hematologic Malignancies
Keywords: Hematologic Neoplasms; Blood Disorders; Blood Cancer; Transplantation, Blood And Marrow; Acute myelogenous leukemia; Myelodysplastic syndrome; Acute lymphocytic leukemia; Aplastic anemia; Chronic myelogenous leukemia; Chronic lymphocytic leukemia; Myeloproliferative disease; Hodgkin's disease; Non-Hodgkin's lymphoma; Multiple myeloma; Cyclophosphamide; Fludarabine; Melphalan; Mesna; Rituximab; Tacrolimus; Prograf; Mycofenolate mofetil; MMF; CellCept; G-CSF; Filgrastim; Neupogen
MeSH Terms: conditions — Leukemia; Hematologic Neoplasms; Hematologic Diseases; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Aplastic; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myeloproliferative Disorders; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Melphalan; Mesna; Rituximab; Stem Cell Transplantation; Thiotepa; Tacrolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Haploidentical related (Experimental): Arm 1 - Stem Cell Transplantation (SCT), Melphalan 140 mg/m^2 , Thiotepa 5 mg/kg, Fludarabine 40 mg/m^2 + high-dose post-transplant cyclophosphamide 50 mg/kg/day
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Melphalan; Drug: Mesna; Drug: Rituximab; Procedure: Stem Cell Transplantation; Drug: Thiotepa; Drug: Tacrolimus; Drug: Mycofenolate mofetil; Drug: G-CSF
- 1 Antigen Mismatch Related or Unrelated (Experimental): Arm 2 - SCT, Melphalan, Thiotepa, Fludarabine + high-dose post-transplant cyclophosphamide.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Melphalan; Drug: Mesna; Drug: Rituximab; Procedure: Stem Cell Transplantation; Drug: Thiotepa; Drug: Tacrolimus; Drug: Mycofenolate mofetil; Drug: G-CSF
- Matched Unrelated Donor (MUD) (Experimental): Arm 3 - SCT, Melphalan, Thiotepa, Fludarabine + high-dose post-transplant cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Melphalan; Drug: Mesna; Drug: Tacrolimus; Drug: Mycofenolate mofetil; Drug: G-CSF

INTERVENTIONS:
Drug: Cyclophosphamide — 50 mg/kg/day intravenous (IV) over 3 hours on Days 3 and 4.
  Other Names: Cytoxan; Neosar
Drug: Fludarabine — 40 mg/m^2 IV over 1 hour on Days -6, -5, -4, and -3.
  Other Names: Fludara; Fludarabine Phosphate
Drug: Melphalan — 140 mg/m^2 IV (or 100 mg/m^2 with reduced intensity Regimen 2) over 30 minutes on Day -8.
  Other Names: Alkeran
Drug: Mesna — 10 mg/kg IV every 4 hours for a total of 10 doses starting just prior to first dose of Cyclophosphamide on Days 3 and 4.
  Other Names: Mesnex
Drug: Rituximab — CD20+ lymphoid malignancies: 375 mg/m2 on Day -13 followed by 1000 mg/m2 on Day -6, +1, and +8.
  Other Names: Rituxan
  Arms: 1 Antigen Mismatch Related or Unrelated; Haploidentical related
Procedure: Stem Cell Transplantation — Infusion of donor's stem cells by vein on Day 0, may last anywhere from 15 minutes to several hours.
  Other Names: SCT; Blood Marrow Transplantation; Allogeneic stem cell transplantation; ASCT
  Arms: 1 Antigen Mismatch Related or Unrelated; Haploidentical related
Drug: Thiotepa — 5 mg/kg Regimen 1 (or 5 mg/kg with reduced intensity Regimen 2) IV over 4 hours on Day -7.
  Arms: 1 Antigen Mismatch Related or Unrelated; Haploidentical related
Drug: Tacrolimus — 0.015 mg/kg by vein or orally daily starting on Day +5 for 3 months
  Other Names: Prograf
Drug: Mycofenolate mofetil — 15 mg/kg/dose orally three times a day starting on Day +5 to Day +100 or otherwise indicated
  Other Names: MMF; CellCept
Drug: G-CSF — 5 mcg/kg/day subcutaneously starting Day 7 once a day daily until neutrophil recovery > 1000/mcl.
  Other Names: Filgrastim; Neupogen

SUMMARY:
The goal of this clinical research study is to learn about the safety of giving a stem cell transplant from a tissue-mismatched donor, followed by cyclophosphamide, to patients with certain types of blood disorders or blood cancers. Melphalan, thiotepa, and fludarabine will also be given before the transplant.

Researchers will study the health status of these patients at 3 months after the transplant.

DETAILED DESCRIPTION:
The Study Treatment:

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

In this study, researchers want to learn if cyclophosphamide can help to prevent graft-versus-host disease (GVHD -- when transplanted immune tissue, such as white blood cells, attacks the tissues of the recipient's body).

Melphalan, thiotepa, and fludarabine are commonly used in combination with a stem cell transplant.

Study Treatment Administration:

If you are found to be eligible to take part in this study, you will receive chemotherapy for 6 days:

* You will receive melphalan by vein over 30 minutes on Day -8 (8 days before the transplant).
* You will receive thiotepa by vein over 4 hours on Day -7.
* You will receive fludarabine by vein over 1 hour on Days -6, -5, -4, and -3.

If thiotepa is not available, you will receive melphalan by vein over 30 minutes on Day -6 and fludarabine by vein over 1 hour on Days -5, -4, -3, and -2. You will receive total body irradiation (TBI) on Day -1.

On Day 0, you will receive the donor's stem cells by vein. This may last anywhere from 15 minutes to several hours.

On Days 3 and 4, you will receive cyclophosphamide by vein over 3 hours. You will also receive mesna by vein over 30 minutes every 4 hours for a total of 10 mesna doses on Days 3 and 4. Mesna is given to lower the risk of side effects to the bladder.

Starting on Day 5, you will receive tacrolimus and mycophenolate mofetil (MMF) to help lower the risk of GVHD. Tacrolimus will be given by vein as a continuous infusion for about 2 weeks. After the 2 weeks of taking tacrolimus by vein, you will take tacrolimus by mouth as a pill for at least 3 months. MMF will be given by mouth, 3 times a day, usually until Day 35.

Starting on Day 7, you will receive filgrastim (G-CSF) once a day as an injection under the skin, until your blood cell counts reach a high enough level.

Depending on the type of disease that you have, your doctor may decide to give you rituximab by vein over several hours on Days -13, -6, 1, and 8. Rituximab is given to help the body get rid of abnormal white blood cells.

Length of Study Participation:

You will be in the hospital for about 4 weeks after the transplant. You will be taken off study if the disease gets worse. The study drugs will be stopped if intolerable side effects occur.

Follow-Up Visits:

You will be asked to stay close enough to Houston to be able to come back for any visits for at least 100 days after the transplant.

At 1, 3, 6, and 12 months after the transplant, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 4 tablespoons) will be drawn for routine tests.
* You will have a bone marrow biopsy/aspirate to check the status of the disease. If you have lymphoma or aplastic anemia, you may have a bone marrow biopsy/aspirate at 3, 6, and 12 months, if your doctor thinks it is needed.
* Blood (about 4 tablespoons) will be drawn to measure tumor cells and to predict graft failure and/or relapse.
* You may have urine collected and/or scans performed such as x-rays, CT scans, and/or a positron emission tomography (PET) scan. These scans and urine tests would only be done if the study doctor thinks they are needed to check the status of the disease.
* Blood (about 4 tablespoons) will be drawn to check your immune system.

If you have AML, at 2 months after the transplant, blood (about 4 tablespoons) will be drawn to check your immune system.

If you have MM, you will have a bone survey once a year.

If the study doctor thinks it is needed based on side effects you may be having, additional follow-up tests will be performed.

You may be contacted by phone 1-2 times a year to ask about the status of the disease. These calls will take about 10 minutes to complete.

This is an investigational study. All of the drugs used in this study are commercially available and FDA approved. However, it is investigational to give high-dose cyclophosphamide for preventing GVHD that may occur after a stem cell transplant from a tissue-mismatched donor.

Up to 337 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients < 55 years (Myeloablative regimen #1) or > 55 and </= 75 years or significant comorbidities (Reduced intensity regimen #2) old lacking a matched related volunteer donor identified in time for transplant for which a related haploidentical donor (</= 7/8 allele match at the A, B, C, DR loci), a 7/8 allele matched related or unrelated donor is identified, or a matched unrelated donor (MUD). The patients must be diagnosed with a high-risk disease defined as following:
2. Acute lymphocytic leukemia (ALL) in CR1 with high-risk features including adverse cytogenetics such as t(9;22), t(1;19), t(4;11), or MLL gene rearrangements; ALL in second or greater remission or ALL with relapsed disease, peripheral blood blasts < 1000/microliter, ALL patients must show response to most recent received chemotherapy;
3. Acute myeloid leukemia (AML) in CR1 with intermediate-risk disease or high-risk features defined as: Greater than 1 cycle of induction therapy required to achieve remission; Preceding myelodysplastic syndrome (MDS) or myeloproliferative disease; Presence of FLT3 mutations or internal tandem duplications; FAB M6 or M7 classification; Adverse cytogenetics, -5, del 5q, -7, del7q, abnormalities involving 3q, 9q, 11q, 20q, 21q, 17, +8 [> 3 abnormalities], peripheral blood blasts <1000/microliter, AML patients must show response to most recent received chemotherapy;
4. AML in second or greater remission, primary induction failure and patients with relapsed disease, peripheral blood blasts <1000/microliter; patients > 55 years and </= 75 years need to be in morphologic remission at transplant (< 5% blasts).
5. Myelodysplastic syndrome (MDS) with International Prognostic Scoring System (IPSS) intermediate-2 or higher; or therapy-related MDS
6. Aplastic anemia with Absolute neutrophil count (ANC)<1000 and transfusion dependent after they failed immunosuppression therapy
7. Chronic myeloid leukemia (CML) >/=1st chronic phase, after failed >/=2 lines of tyrosine kinase inhibitors; in accelerated or blast phase with > 30% bone marrow blasts;
8. Prior allogeneic stem cell transplant more than 6 months from the first transplant, in remission.
9. Chemotherapy-sensitive relapsed lymphoma (Complete or partial response), Hodgkin's or non-Hodgkin's lymphoma, no evidence of "bulky" disease (> 10 cm in diameter);
10. Patients with chemo-sensitive CLL with persistent or recurrent disease after fludarabine-based regimens, no evidence of "bulky" disease (> 10 cm in diameter)
11. Patients with poor prognosis multiple myeloma by cytogenetics (del13, del 17p, t(1;14) or t(14;16) or hypodiploidy, with advanced disease (stage>/=2) and /or relapsed after autologous stem cell transplant.
12. Patients with myelofibrosis (Lille >0, transfusion dependency, progression to blast phase; however, in remission from AML) or chronic myelomonocytic leukemia (CMML). These patients will be treated with the reduced-intensity conditioning regimen #2 and will be subject to the same stopping rule as the group >/= 55 years or with comorbidities.
13. Zubrod performance status 0-1 or Lansky PS greater or equal to 70%.
14. Patients above >/=65 years old should have an age-adjusted co-morbidity index of </= 3.
15. Available donor able to undergo a bone marrow harvest. For matched unrelated donor transplants only: Peripheral blood stem cells may be collected if donor is unavailable for bone marrow harvest or if adequate bone marrow cannot be collected.
16. Bilirubin </= 1.5 mg/dl (unless Gilbert's syndrome), ALT or AST </= 200 IU/ml.
17. Serum creatinine clearance >/=50 ml/min (calculated with Cockcroft-Gault formula); Creatinine for children </=1.5 mg/dl or </=2 times upper limit of normal for age (whichever is less);
18. Diffusing capacity for carbon monoxide (DLCO) >/= 45% predicted corrected for hemoglobin. For pediatric patients, if unable to perform pulmonary function, >/= 92% oxygen saturation with pulse oximetry.
19. Left ventricular ejection fraction (LVEF) >/= 40%.
20. Patient or patient's legal representative, parent(s) or guardian should provide written informed consent. Assent of a minor if participant's age is at least seven and less than eighteen years.

Exclusion Criteria:

1. HIV positive; active hepatitis B or C
2. Patients with active infections. The PI is the final arbiter of the eligibility.
3. Liver cirrhosis with greater than grade 1 stage 1 inflammation/fibrosis
4. Uncontrolled central nervous system (CNS) involvement by tumor cells
5. Patients with AML must have less than 30% bone marrow blasts and no peripheral blood blasts.
6. History of another primary malignancy that has not been in remission for at least 3 years. (The following are exempt from the 3-year limit: non-invasive nonmelanoma skin cancer, fully excised melanoma in situ [Stage 0], curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear.)
7. Positive Beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
8. Inability to comply with medical therapy or follow-up.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-11-05 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Ciurea, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled during the period from January 2010 through August 2014 and were assigned to the HAPLO arm or the 9/10 MUD arm based on donor availability and physician preference. The 3 arms received identical melphalan-based conditioning chemotherapy and GVHD prophylaxis
Pre-assignment Details: Additional arm elderly patients did not accrue any participants so therefore was excluded from summary.
Groups:
- Haplo Arm: Patients that received a stem cell transplant from a haploidentical donor.
- 1AgMM Related/Unrelated Donors: Patients that received a transplant from a 1 antigen mismatched related or unrelated donor
- MUD Donor: Patients that received a transplant from a matched unrelated donor
- Second Transplant: Patients receiving a second transplant
- Myelofibrosis: Patients with the diagnosis of Myelofibrosis
Period: Overall Study
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Started | 89 | 56 | 22 | 6 | 3
Completed | 84 | 51 | 21 | 0 | 0
Not Completed | 5 | 5 | 1 | 6 | 3
Not completed — Lost to Follow-up | 4 | 5 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Haplo Arm: Patients that received a transplant from a haploindentical donor
- Total: Total of all reporting groups
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis | Total
Number analyzed (Participants) | 84 | 51 | 21 | 6 | 3 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 0 | 0 | 0 | 3
  Between 18 and 65 years | 79 | 48 | 11 | 6 | 3 | 147
  >=65 years | 3 | 2 | 10 | 0 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 25 | 6 | 1 | 1 | 75
  Male | 42 | 26 | 15 | 5 | 2 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 1 | 0 | 1 | 0 | 12
  Not Hispanic or Latino | 69 | 46 | 20 | 3 | 3 | 141
  Unknown or Not Reported | 5 | 4 | 1 | 2 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 4 | 0 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 7 | 0 | 0 | 2 | 31
  White | 50 | 36 | 20 | 4 | 1 | 111
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 1 | 2 | 0 | 12
Patients with hematologic malignancies without a matched donor [Count of Participants; unit: Participants] | 84 | 51 | 21 | 6 | 3 | 165

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-relapse Mortality (NRM)
Description: Non-relapse mortality (NRM) is defined as death from any cause other than relapse disease. Bayesian monitoring scheme described in Thall, Simon, and Estey (1996) employed to perform interim monitoring of the data during the course of the trial separately within each group.
Time Frame: At 100 days
Population: Second Transplant and Myelofibrosis was not evaluated due to low accrual.
Measure: Count of Participants; unit: Participants
Groups:
- Haplo Arm: Patients that received a transplant from a haploidentical donor
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Number analyzed (Participants) | 84 | 51 | 21 | 0 | 0
Participants | 8 | 7 | 2 | 0 | 0

2. Secondary Outcome: Number of Participants With Non Related Mortality (NRM)
Description: Non-relapse mortality (NRM) is defined as death from any cause other than relapse disease.
Time Frame: six months
Population: Second Transplant and Myelofibrosis was not evaluated due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Number analyzed (Participants) | 84 | 51 | 21 | 0 | 0
Participants | 17 | 15 | 4 | 0 | 0

3. Secondary Outcome: Engraftments
Time Frame: Day 28
Population: Second Transplant and Myelofibrosis was not evaluated due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Number analyzed (Participants) | 84 | 51 | 21 | 0 | 0
Participants | 80 | 50 | 21 | 0 | 0

4. Secondary Outcome: Grade III-IV aGVHD
Description: Acute Graft vs host disease
Time Frame: 100 days
Population: Second Transplant and Myelofibrosis was not evaluated due to low accrual
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Number analyzed (Participants) | 84 | 51 | 21 | 0 | 0
Participants | 11 | 7 | 1 | 0 | 0

5. Secondary Outcome: cGVHD
Description: Chronic graft vs host disease
Time Frame: 1 year
Population: Second Transplant and Myelofibrosis was not evaluated due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Number analyzed (Participants) | 84 | 51 | 21 | 0 | 0
Participants | 11 | 7 | 0 | 0 | 0

6. Secondary Outcome: Disease Free Survival
Description: Participants who have survived without their original disease.
Time Frame: 1 year
Population: Second Transplant and Myelofibrosis was not evaluated due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
Number analyzed (Participants) | 84 | 51 | 21 | 0 | 0
Participants | 50 | 24 | 12 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the preparative regiment up to day 100.
Arm/Group | Haplo Arm | 1AgMM Related/Unrelated Donors | MUD Donor | Second Transplant | Myelofibrosis
All-Cause Mortality (participants affected / at risk) | 22/84 | 21/51 | 9/21 | 2/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 8/84 | 11/51 | 7/21 | 2/6 | 2/3
Other Adverse Events (participants affected / at risk) | 84/84 | 51/51 | 21/21 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Haplo Arm (N=84) | 1AgMM Related/Unrelated Donors (N=51) | MUD Donor (N=21) | Second Transplant (N=6) | Myelofibrosis (N=3)
Acute renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Adenocirus viremia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Altered mental status (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
BK virus associated hemorrhagic cystitis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 3 | 0 | 0 | 0 | 0
Chronic GI GVHD (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
GI GVHD (Gastrointestinal disorders) | 2 | 4 | 2 | 0 | 0
Headache (General disorders) | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 2 | 2 | 1 | 2 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 1 | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Fungal pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Graft failure (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper GI GVHD (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Haplo Arm (N=84) | 1AgMM Related/Unrelated Donors (N=51) | MUD Donor (N=21) | Second Transplant (N=6) | Myelofibrosis (N=3)
Acute renal failure (Renal and urinary disorders) | 4 | 5 | 3 | 0 | 1
Altered mental status (Nervous system disorders) | 4 | 3 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
BK virus associated hemorrhagic cystitis (Renal and urinary disorders) | 37 | 18 | 6 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
C difficile colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 3 | 3 | 2 | 1 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0
Chemo Burn (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Chorioretinitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic GI GVHD (Gastrointestinal disorders) | 4 | 3 | 0 | 0 | 0
Chronic Liver GVHD (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Chronic Ocular GVHD (Eye disorders) | 1 | 0 | 0 | 1 | 0
Chronic Oral GVHD (General disorders) | 3 | 0 | 0 | 0 | 0
Chronic Skin GVHD (Skin and subcutaneous tissue disorders) | 7 | 2 | 0 | 0 | 0
CMV chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DAH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Delayed Engraftment (Blood and lymphatic system disorders) | 3 | 3 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 55 | 33 | 15 | 4 | 1
Disseminated toxoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Elevated ALK Phosphatase (Hepatobiliary disorders) | 7 | 5 | 3 | 0 | 0
Elevated ALT (Hepatobiliary disorders) | 19 | 12 | 5 | 3 | 0
Elevated AST (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Elevated bilirubin (Hepatobiliary disorders) | 21 | 20 | 3 | 1 | 2
Elevated WBC (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Endocarditis (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Fever (Investigations) | 13 | 5 | 2 | 1 | 0
Fluid overload (Investigations) | 61 | 29 | 18 | 5 | 3
GI bleed (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
GI GVHD (Gastrointestinal disorders) | 14 | 9 | 6 | 2 | 2
GI pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Hand/Foot syndrome (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 0
Headache (General disorders) | 8 | 2 | 0 | 0 | 0
Hemorrhagic cystitis (Renal and urinary disorders) | 5 | 4 | 1 | 0 | 1
Hypertension (Cardiac disorders) | 18 | 19 | 5 | 0 | 2
Idiopathic pneumonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 65 | 38 | 19 | 2 | 2
Fungal infection (Infections and infestations) | 5 | 6 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 70 | 36 | 17 | 5 | 3
Liver GVHD (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 1
Metabolic encephalopathy (General disorders) | 0 | 3 | 0 | 0 | 0
Mucositis (Gastrointestinal disorders) | 41 | 30 | 9 | 4 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 84 | 51 | 21 | 6 | 2
Neutropenic fever (Infections and infestations) | 38 | 16 | 1 | 2 | 2
Neutropenic Typhlitis (Infections and infestations) | 1 | 2 | 1 | 0 | 1
Orthostatic hypotension (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 | 5 | 8 | 0 | 0
Fungal pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1 | 0 | 0
HSV oral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Graft failure (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Skin rash (Skin and subcutaneous tissue disorders) | 5 | 7 | 1 | 0 | 0
Renal insufficiency (Renal and urinary disorders) | 11 | 5 | 2 | 2 | 3
Secondary graft failure (Blood and lymphatic system disorders) | 11 | 0 | 3 | 1 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
Skin GVHD (Skin and subcutaneous tissue disorders) | 21 | 17 | 6 | 4 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 1 | 0 | 0
Infusion reaction (Investigations) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0 | 0
Tremors (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
TMA (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0
Upper GI GVHD (Gastrointestinal disorders) | 26 | 11 | 8 | 3 | 1
Veno occlusive disease (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT01010217/Prot_SAP_000.pdf